CLINICAL TRIAL: NCT06135844
Title: Herpes Simplex Virus-1: A Pilot Study Using Hand Sanitizer
Brief Title: Hand Sanitizer Use for Herpes Simplex Virus-1
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leciel Bono (Other)
Responsible Party: Sponsor-Investigator, Leciel Bono, Associate Professor, Graduate Program Director/Interim Dept. Chair, Idaho State University
Organization: Idaho State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-172
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Virus; HSV-1; Herpes Simplex 1; Herpes Simplex Labialis
Keywords: Virus; HSV-1; Herpes Simplex 1; Herpes Simplex Labialis
MeSH Terms: conditions — Virus Diseases; Herpes Labialis | interventions — Hand Sanitizers; Mineral Oil

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups: Control Group (mineral oil) and the Treatment Group (hand sanitizer). Each group will be asked to apply the product to the HSV-1 lesion. Sample Inclusion Criteria: For the purpose of this study participants must be in the early prodromal stage of an HSV-1 outbreak (less than 24 hours from initial symptom), with the visible manifestation of a lesion, 18 years or older, capable of following daily treatment instructions, willing to complete a daily journal and willing to come to either clinic twice for photos during the duration of the lesion (day 3 and when the lesion has healed or the crust has fallen off the lesion).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Hand Sanitizer) (Experimental): Participants with an early prodromal stage of an HSV-1 outbreak (less than 24 hours from initial symptom), with the visible manifestation of a lesion will be invited to participate in the study. Participants will apply a large drop of hand sanitizer in an unmarked container to a Q-tip and will hold the Q-tip on the lesion for 10 seconds. The hand sanitizer will be administered every waking hour in the same manner.
  Interventions: Drug: Purell Hand Sanitizer
- Control Group (Medical Grade Mineral Oil) (Placebo Comparator): Participants with an early prodromal stage of an HSV-1 outbreak (less than 24 hours from initial symptom), with the visible manifestation of a lesion will be invited to participate in the study. Participants will apply a large drop of Medical Grade Mineral Oil in an unmarked container to a Q-tip and will hold the Q-tip on the HSV-1 lesion for 10 seconds. The medical grade mineral oil will be administered every waking hour in the same manner.
  Interventions: Drug: Medical Grade Mineral Oil

INTERVENTIONS:
Drug: Purell Hand Sanitizer — Active ingredient. Ethyl alcohol 70%
  Other Names: Hand Sanitizer
  Arms: Treatment Group (Hand Sanitizer)
Drug: Medical Grade Mineral Oil — Inert ingredients: Saturated hydrocarbons, with a purity and chemical structure that differs substantially from food-grade or technical-/industrial-grade mineral oils.
  Other Names: Mineral Oil
  Arms: Control Group (Medical Grade Mineral Oil)

SUMMARY:
The purpose of this pilot study is to determine if the use of Purell hand sanitizer alters the duration, level of pain and discomfort during treatment, and the size of the HSV-1 lesion. The duration of an HSV-1 (herpes) lesion is the primary endpoint for this study. Size, pain, and discomfort are the secondary endpoints.

DETAILED DESCRIPTION:
The participants will be divided into a control group (10 participants) and treatment group (10 participants) and will be given either the Purell hand sanitizer (treatment group) or medical grade mineral oil (control group) to treat the lesion. Participants will apply a large drop of the product (purell hand sanitizer or mineral oil) on a q-tip and will hold the q-tip on the lesion for 10 seconds. Participants will be instructed to apply a solution to lesion every waking hour for the next 14 days or until lesion has healed. Each day the participant will fill out the daily journal. The journal includes a measurement in millimeters of the lesion with graph paper, recorded number of applications for that day, and two visual analog scales- one measuring any discomfort from the lesion and the other recording the pain during the application process.

Documentation of changes to the lesion will be recorded in a daily journal until the lesion is healed. There are two days that the participants are expected to return to the clinic for re-examination at day three and the last day when the lesion has healed, or the crust has fallen off. Pictures of the lesion will taken at these two points in time.

The duration the HSV-1 lesion, level of pain and discomfort during treatment, and the size of the HSV-1 lesion will be statistically measured between the control group (mineral oil) and the treatment group (purell hand sanitizer) to determine if there is any statistical difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

For the purpose of this study participants must be:

* in the early prodromal stage of an HSV-1 outbreak (less than 24 hours from initial symptom)
* have a visible manifestation of a lesion
* be 18 years or older
* capable of following daily treatment instructions
* willing to complete a daily journal
* willing to come to the clinic twice for records and pictures during the14 days that the lesion is present or until participant is free of lesion.

Exclusion Criteria:

For the purpose of this study participants cannot:

* be immunocompromised
* be pregnant
* have taken any antiviral medication within the last two weeks
* have used any creams in the last ten days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Duration of HSV-1 Lesion | 1-14 days
  1. Is there a statistically significant difference in the duration of the HSV-1 lesion in individuals who use Purell hand sanitizer on their lesion versus those who are in the control group using medical grade mineral oil? The duration will be determined when the crust of the lesion has fallen off and the lesion is fully healed. Once healed, the participant will be required to return to the clinic for a concluding photograph taken by the research assistant and return the daily journal.

SECONDARY OUTCOMES:
Level of Pain during Treatment | 1-14 days
  2. Is there a statistically significant difference in the level of pain during the treatment application process of an HSV-1 lesion for those who use Purell hand sanitizer on their lesion versus those who are in the control group using medical grade mineral oil? Pain will be measured by the participants daily using a Visual Analog Scale (VAS) which ranges from 1-10 with 1=no pain and 10=extreme pain. The higher the score in the VAS scale, the more pain the participant is experiencing. The pain scale will be used after the medication is applied to determine if there is any corresponding pain with the medication.
Level of Discomfort during Treatment | 1-14 days
  Is there a statistically significant difference in the level of discomfort during an HSV-1 lesion for those who use Purell hand sanitizer on their lesion versus those who are in the control group using medical grade mineral oil? Level of discomfort will be measured by the participants daily using a Visual Analog Scale (VAS) which ranges from 1-10 with 1=no pain and 10=extreme pain. The higher the score the VAS scale, the higher the level of discomfort with the HSV-1 lesion. The level of discomfort refers to the overall discomfort from the lesion experienced by participants on that day.
Size of Lesion during Treatment | 1-14 days
  Is there a statistically significant difference in the size of the HSV-1 lesion for those who use Purell hand sanitizer on their lesion versus those who are in the control group using medical grade mineral oil? The size of the lesion will be measured daily by the participant using millimeter markings on a laminated ruler provided in the kit. Participants will be given instructions on how to measure the lesion using this ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Leciel Bono, MS, Study Chair — Idaho State University
Locations (3):
- United States (3):
  - Idaho State University, Pocatello, Idaho
  - Cotton Creek Dental, St. George, Utah
  - Utah Tech University, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angewandte V. As a biocidal active substance, ethanol is indispensable for hygienic hand disinfection. Zentralsterilisation. 2020; 28(6):354-359. Our study has never been investigated by researchers. This is a pilot study exploring the effectiveness of ethyl alcohol on HSV-1 lesions. Therefore all research studies pertain to the virucidal effects of 70% ethyl alcohol.
- [Background] Sauerbrei A. Bactericidal and virucidal activity of ethanol and povidone-iodine. Microbiologyopen. 2020 Sep;9(9):e1097. doi: 10.1002/mbo3.1097. Epub 2020 Jun 22. PMID 32567807
- See also: World Health Organization. Guideline on Hand Hygiene in Healthcare. 2009. — http://apps.who.int/iris/bitstream/handle/10665/44102/9789241597906_eng.pdf
- See also: U.S. Food and Drug Administration (2019, April 11). If soap and water are not available, hand sanitizers may be a good alternative. — http://www.fda.gov/consumers/if-soap-and-water-are-not-available-hand-sanitizers-may-be-good-alternative